CLINICAL TRIAL: NCT02957955
Title: Cardiovascular Prehabilitation in Patients Awaiting Heart Transplantation - Addressing Clinical Needs (PREHAB HTx Study)
Brief Title: Cardiovascular Prehabilitation in Patients Awaiting Heart Transplantation (PREHAB HTx Study)
Acronym: PREHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20160753-01H
Record Dates: First submitted 2016-10-27; First posted 2016-11-08 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure
Keywords: Heart failure
MeSH Terms: conditions — Heart Failure | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Group 1. Usual care + High-Intensity Interval Training, Nutritional Workshop, Stress Management Course.
  Interventions: Behavioral: High-Intensity Interval Training
- Non interventional (No Intervention): Group 2. Usual care. Patients are encouraged to remain physically active, although they do not participate in a regular structured exercise training program.

INTERVENTIONS:
Behavioral: High-Intensity Interval Training — Participants will complete supervised exercise sessions. Participants will attend on-site high-intensity interval training two times weekly for 12 weeks. Participants will complete six-minute walk test, cardiopulmonary exercise test, and six questionnaires: Short Form 36 Health Survey Questionnaire (SF-36), Minnesota Living with Heart Failure Questionnaire (MLHFQ), Beck Depression Inventory II (BDI-II), Beck Anxiety Inventory (BAI), Montreal Cognitive Assessment (MOCA), and Impact of Events Scale-Revised (IES-R) at baseline (week 1) and follow-up (after 12 weeks of intervention).
  Arms: Interventional

SUMMARY:
This study evaluates the addition of high-intensity interval training to the standard pre-heart transplantation clinical care. Participants will be randomised into 2 arms: one arm will receive high-intensity interval training, and the other arm will be encouraged to remain physically active, although they do not participate in a regular structured exercise training program.

DETAILED DESCRIPTION:
Heart failure affects more than 6.2 million people living in North America. Approximately 10% of patients with heart failure have advanced heart failure. Heart transplantation is an effective life-saving treatment for patients with advanced heart failure. The cardiovascular rehabilitation programs are integral to heart failure management.

This study is being done to evaluate, in adults with advanced heart failure awaiting heart transplantation, the effects of cardiovascular rehabilitation (including high-intensity interval training, stress management and nutrition workshops) on functional capacity, aerobic power, frailty, quality of life, and mental health.

This study compares pre-transplant cardiovascular rehabilitation with usual pre-transplant care in patients with advanced heart failure awaiting heart transplant.

All participants will be randomized into 2 study groups: Group 1 (rehab), and Group 2 (no rehab). Those randomized to Group 1 will receive usual care, 12 weeks of rehab (exercise training, and attend stress and nutrition course through the Heart Failure Clinic and the Division of Prevention and Rehabilitation at the University of Ottawa Heart Institute). Those randomized to Group 2 will receive regular visits through the Heart Failure Clinic; patients are encouraged to remain physically active, although they do not participate in a regular structured exercise training program.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced heart failure and listed for heart transplantation.
2. Able to perform a symptom-limited exercise test.
3. Age =>18 years old.
4. Able to provide informed consent.

Exclusion Criteria:

1. Currently participating in a structured exercise training program (> 2 times per week)
2. Status 4 priority listing for heart transplantation.
3. Myocardial infarction =<7 days.
4. Heart failure with hemodynamic instability.
5. Hypertrophic obstructive cardiomyopathy with symptomatic left ventricular outflow tract gradient =>30 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-02-02 (Actual)

PRIMARY OUTCOMES:
Change in functional capacity | Baseline to 12 weeks
  Change in in functional capacity from baseline to 12 weeks as measured by six-minute walk test distance. Distance walked will be measured in meters.

SECONDARY OUTCOMES:
Change in aerobic power | Baseline to 12 weeks
  Measured using expired VO2 gas samples, measured in L/min, ml/kg/min
Change in frailty | Baseline to 12 weeks
  Measured by the Fried criteria. Measured by presence of 3 out of 5 frailty symptoms.
Change in general quality of life | Baseline to 12 weeks
  Measured by the Short Form 36 Health Survey Questionnaire (SF-36). The SF-36 consists of 8-scaled scores which are the weighted sums of the questions in their section.
Change in disease-specific quality of life | Baseline to 12 weeks
  Measured by the Minnesota Living with Heart Failure Questionnaire (MLHFQ). MLHFQ is a 21-item scale that measures the effects of heart failure on quality of life using a 6-point scale.
Change in depressive symptoms | Baseline to 12 weeks
  Measured by the Beck Depression Inventory II (BDI-II). It contains 21-questions, each answer being scored on a scale of 0 to 3.
Change in anxiety | Baseline to 12 weeks
  Measured by the Beck Anxiety Inventory (BAI). The BAI is a 21-item validated self-reported measure. A total score is calculated by summing the items; maximum score is 62.
Change in cognitive function | Baseline to 12 weeks
  Measured by the Montreal Cognitive Assessment (MOCA). The MOCA is made up of 8 subscales, scores are totaled; maximum score is 30 points.
Change in response to a specific traumatic event | Baseline to 12 weeks
  Measured by the Impact of Events Scale- Revised (IES-R). IES-R is 22 items, zero to four scale. Scores above 23 are of concern; scores above 32 indicate a probable diagnosis of PTSD.
Short term post-heart transplantation outcomes | One year post-heart transplantation
  Data collected from medical records: length of hospital stay, adverse events (infection, treated rejection, bleeding, and stroke), survival to hospital discharge, and 30 day hospital readmissions.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Reed, Ph.D, R.Kin, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (2):
- Canada (2):
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Reed JL, Tulloch HE, Ross H, Terada T, Mistura M, Marcal IR, Oh P, Chih S. Cardiovascular Prehabilitation in Patients Awaiting Heart Transplantation- Addressing Clinical Needs (the PREHAB HTx Study). CJC Open. 2025 May 22;7(8):1110-1119. doi: 10.1016/j.cjco.2025.05.009. eCollection 2025 Aug. PMID 40894839